CLINICAL TRIAL: NCT03253575
Title: CANscriptTM Clinical Outcomes in a Real-World Setting (ANCERS)-2: A Prospective, Multicenter, Observational Study Examining the Clinical Utility of CANscriptTM in Routine Clinical Practice
Brief Title: CANscriptTM Clinical Outcomes in a Real-World Setting (ANCERS)-2
Acronym: ANCERS-2
Status: Suspended | Type: Observational
Why Stopped: Mitra is temporarily suspending enrollment in the ANCERS-2 clinical utility study due to unexpected test performance results, to analyze the test performance.
Sponsor: Mitra RxDx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MIT-201701
Record Dates: First submitted 2017-08-09; First posted 2017-08-18 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2018-12

CONDITIONS: Adult Solid Tumor
Keywords: Head and Neck Squamous Cell Carcinoma; Breast Cancer; Non-Small Cell Lung Cancer; Epithelial Ovarian Cancer; Colorectal Cancer; Local Recurrent Cancer; Late Stage Cancer; Clinical Utility; Outcomes Study
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue biopsies and resections embedded formalin fixed paraffin and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Squamous Carcinoma of the Head and Neck (HNSCC): 1st line metastatic/locally advanced
  * 2nd line metastatic/locally advanced
  Interventions: Diagnostic Test: CANscript
- Triple Negative Breast Cancer (TNBC): 1. Triple Negative Breast Cancer (TNBC) A 1st line metastatic/locally advanced B ≥2nd line metastatic/locally advanced
  Interventions: Diagnostic Test: CANscript
- Non-small Cell Lung Cancer (NSCLC): 1. Non-small Cell Lung Cancer (NSCLC) A ≥2nd line Stage 3B or 4
  Interventions: Diagnostic Test: CANscript
- Epithelial Ovarian Cancer (EOC): 1. Epithelial Ovarian Cancer (EOC) A 2nd line platinum-resistant Stage 3 or 4 B 2nd line platinum-sensitive Stage 3 or 4 C ≥3rd line platinum-sensitive Stage 3 or 4
  Interventions: Diagnostic Test: CANscript
- Colorectal Cancer (CRC): 1. Colorectal Cancer (CRC) A 1st line Stage 4 B Recurrent or progressive disease following treatment with both oxaliplatin- and irinotecan-containing regimens
  Interventions: Diagnostic Test: CANscript

INTERVENTIONS:
Diagnostic Test: CANscript — CANscript is a predictive test that supports informed selection of cancer therapeutics for each individual patient. CANscript has the potential to predict the response of the patient under evaluation to either single-agent cancer therapeutics or combination therapeutic regimens. This is accomplished by using fresh tumor tissue from the patient in plates coated with a specific set of tumor matrix proteins (TMP). Further, patient derived autologous ligands are added to the culture. Angiogenic factors are added to maintain tumor vasculature along with autologous immune cells. In essence, CANscript recapitulates the tumor microenvironment.

SUMMARY:
The purpose of this study is to test the CANscript™ sensitivity assay, which is a new and different assay developed to test the sensitivity of different cancer types to physician selected therapies (both drugs and/or drug combinations) indicated for the stage and type of cancer for treatment. CANscript™ tests how a patients specific tumor reacts to the therapies being considered by the treating physician. CANscript™ test results have been shown to closely correspond with actual clinical results, providing physicians with information that may help him/her develop a more personalized cancer treatment and care plan based on the patients specific condition. The researchers want to see if CANscript™ test results are helpful in selecting the treatments prescribed and provided. There will be about 800 people taking part in this study, across 5 different tumor types. The study is designed to assess the decision impact of the CANscript™ test results in informing physicians in therapy selection.

DETAILED DESCRIPTION:
This is an observational data collection study evaluating how physicians utilize therapeutic sensitivity information ascertained with CANscript, and subsequently describing clinical outcomes (clinical response and survival) resulting from their therapeutic selection.

Potential patients presenting for study enrollment will provide written informed consent and will subsequently be screened per inclusion/ exclusion criteria. Once enrolled, a biopsy & blood draw will be scheduled to obtain material for CANscript testing. Imaging will also be scheduled if a fresh image (obtained within 14 days of planned treatment initiation) is not available. Prior to submitting a fresh tissue sample for CANscript, the treating physician will select any number of therapies being considered for treatment, and will assign a priority ranking to those therapies (priority #1 through priority #N, with #1 representing their most preferred therapeutic option for the patient, and #N representing the number of their least preferred of the appropriate potential therapies). Prioritized therapies can be either single-agent therapeutics or combination regimens. All ranked therapeutic options must be available for individual patient at the time of selection. The prioritized list of preferred therapies will be sent to the testing laboratory (Mitra Biotech, Inc.) at least 2 days before the biopsy and blood draw are performed. Fresh tumor and blood samples will subsequently be sent to the testing laboratory for receipt within 24 hours of biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥18 years old
2. ECOG performance status of ≤ 2
3. The patient's tumor must be amenable to a tumor biopsy sampling, so that CANscript can be performed
4. The patient must have disease that is measurable by standard imaging techniques, per the RECIST 1.1 (For patients with prior radiation therapy, measurable lesions must be outside of any prior radiation field[s], unless disease progression has been documented at that disease site subsequent to radiation)
5. Histologically- or cytologically-confirmed:

   A Locally advanced or metastatic HNSCC; B Locally advanced or metastatic TNBC; C Locally advanced or metastatic Stage 3b or 4 NSCLC after failure of appropriate 1st line therapy (i) Patients with EGFR or ALK mutations must have received previous appropriate therapy; D Locally advanced or metastatic epithelial ovarian, fallopian tube, or primary peritoneal carcinoma, after failure of 1st line platinum-based chemotherapy (i) Recurrent or persistent stage 3 or 4 disease requiring relapse histologic documentation; E Stage IV metastatic CRC
6. Patient has signed informed consent prior to initiation of any study-specific procedures

Exclusion Criteria:

1. The patient has persistent clinically significant toxicities (Grade ≥2) from previous anticancer therapy (excluding chronic Grade 2 chemotherapy-related neuropathy which is permitted, and excluding Grade 2-3 laboratory abnormalities if they are not associated with symptoms, are not considered clinically significant by the Investigator, and can be managed with available medical therapies).
2. The patient has received treatment with chemotherapy, external-beam radiation, or other systemic anticancer therapy within 14 days prior to study entry (42 days for prior nitrosourea or mitomycin-C). (Patients could have received supportive care therapeutics as appropriate).
3. The patient has an additional active malignancy that may confound the assessment of the study endpoints. Patients with a past cancer history (active malignancy within 2 years prior to study entry) with substantial potential for recurrence must be discussed with the Sponsor before study entry. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia), organ-confined prostate cancer with no evidence of progressive disease.
4. The patient has clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
5. The patient has uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study.
6. The patient has known active or suspected brain or leptomeningeal metastases. (Central nervous system [CNS] imaging is not required prior to study entry unless there is a clinical suspicion of CNS involvement). Patients with stable, treated brain metastases are eligible provided there is no evidence of CNS disease growth on imaging for at least 6 weeks following radiation therapy or other loco-regional ablative therapy to the CNS.
7. The patient is receiving immunosuppressive therapy for prophylaxis following a prior organ transplant (solid organ or allogeneic stem cell). Corticosteroid therapy is permitted.
8. The patient has uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, disseminated intravascular coagulation, or psychiatric illness/social situations that would limit compliance with study requirements.
9. The patient is pregnant or breast-feeding. The patient has known positive status for human immunodeficiency virus active or chronic Hepatitis B or Hepatitis C.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Males or females ≥18 years old, with an ECOG performance status of ≤2 who have recurrent locally advanced or metastatic cancers of the Head and Neck, Colorectal, Triple Negative Breast, Epithelial Ovarian, or Non-Small Cell lung cancers.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-07-13 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
CANscript decision impact will be captured via a study specific questionnaire | 18-24 months
  1. A questionnaire will be used to capture the information to be able to summarize the concordance and discordance rates between:
  1. Empirically selected therapy (selected by treating physicians prior to knowing the CANscript results for a given patient) and CANscript recommended therapy (i.e., the therapy with the highest CANscript M-score for a given patient).
  2. Empirically selected therapy and CANscript results that predict response or non-response.

SECONDARY OUTCOMES:
The RECIST 1.1 criteria will utilized to assess therapy response, i.e. Complete Response (CR), Partial Response (PR), Stable Disease (SD), Duration of Response (DoR), Progression Free Survival (PFS) | 24-48 months
  A baseline Image will be taken prior to therapy initiation, and then as per tratment guidelines throughout and following therapy delivery:
  1. To summarize tumor response in terms of objective response rate (ORR), clinical benefit rate (CBR), duration of response (DoR) progression-free survival (PFS), and overall survival (OS) based on imaging (CT, MRI, etc.) and scoring per RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rowinsky, MD, Study Chair — Chief Medical Officer Mitrabiotech
Locations (30):
- United States (30):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Colorado School of Medicine-Denver, Aurora, Colorado
  - Eastern CT Hematology and Oncology Associates, Norwich, Connecticut
  - Lynn Cancer Institute, Boca Raton, Florida
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Miami-Sylvester Comprehensive Cancer Center, Miami, Florida
  - The Center for Gyencologic Oncology, Miramar, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Tallahassee Memorial Cancer Center, Tallahassee, Florida
  - Memorial Health University Medical Center- Savannah Health Services, Savannah, Georgia
  - Joliet Oncology Associates, Joliet, Illinois
  - Edward Elmhurst Healthcare, Naperville, Illinois
  - Community Hospital, Munster, Indiana
  - Ochsner Health System, New Orleans, Louisiana
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - Michigan Center of Medical Research -MHP, Farmington Hills, Michigan
  - St John Hospital and Medical Center (Great Lakes Cancer Managment Specialists), Grosse Pointe Woods, Michigan
  - War Memorial Hematology/Oncology, Sault Ste. Marie, Michigan
  - Mercy Hospital, St Louis, Missouri
  - University of Rochester/Wilmot Cancer Institute, Rochester, New York
  - Saint Thomas Health, Nashville, Tennessee
  - Austin Cancer Centers, Austin, Texas
  - Doctors Hospital at Renaissance-DHR Health, Edinburg, Texas
  - University of Texas Medical Branch at Galveston(UTMB), Galveston, Texas
  - Oncology Consultants, Houston, Texas
  - Baylor College of Medicine Hemtology/Oncology, Houston, Texas
  - Houston Methodist Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston- Hermann, Houston, Texas
  - Invesclinic US McAllen Oncology, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No